CLINICAL TRIAL: NCT04704895
Title: A Prospective RCT Study of Comparing Early Enteral Nutrition Versus Parenteral Nutrition After Pancreaticoduodenectomy
Brief Title: Comparing Early Enteral Nutrition Versus Parenteral Nutrition After Pancreaticoduodenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xian-Jun Yu (Other)
Responsible Party: Sponsor-Investigator, Xian-Jun Yu, President of Pancreatic Cancer Institute, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CSPAC-32
Record Dates: First submitted 2020-11-28; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Enteral Nutrition
MeSH Terms: interventions — Parenteral Nutrition, Total; Enteral Nutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Total parenteral nutrition (Active Comparator): Total parenteral nutrition, TPN also starts from POD 1 and is delivered through a central venous catheter, with a target energy of 1.5 amino acids/kg/day reaching 30 kcal/kg/day
  Interventions: Dietary Supplement: Total parenteral nutrition
- Arm B: Enteral nutrition (Experimental): NJEEN was defined as providing at least 50% of the nutritional requirements through the nasojejunal tube prior to the 5th day after surgery (POD) and having no parenteral nutrition for 72 hours or more.
  Interventions: Dietary Supplement: Enteral nutrition

INTERVENTIONS:
Dietary Supplement: Total parenteral nutrition — Total parenteral nutrition, TPN also starts from POD 1 and is delivered through a central venous catheter, with a target energy of 1.5 amino acids/kg/day reaching 30 kcal/kg/day
  Arms: Arm A: Total parenteral nutrition
Dietary Supplement: Enteral nutrition — NJEEN was defined as providing at least 50% of the nutritional requirements through the nasojejunal tube prior to the 5th day after surgery (POD) and having no parenteral nutrition for 72 hours or more.
  Arms: Arm B: Enteral nutrition

SUMMARY:
To prove that early enteral nutrition after pancreaticoduodenal operation is of great significance to improve the immune response, reduce the incidence of postoperative infection and other related complications, and shorten the length of hospital stay

DETAILED DESCRIPTION:
Arm A: Total parenteral nutrition. TPN also started from POD 1 and was delivered through a central venous catheter. Target energy of 1.5 amino acids/kg/day reached 30 kcal/kg/day.

Arm B: NJEEN was defined as providing at least 50% of the nutritional requirements through the nasojejunal tube prior to the 5th day after surgery (POD) and having no parenteral nutrition for 72 h or more.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old, gender is not limited;
* All patients underwent pancreaticoduodenectomy;
* ECOG 0 ~ 2 for physical condition score;
* Imaging examination found pancreatic head, periampullary space, no distant metastasis and ascites;
* No bone marrow dysfunction;
* Those without obvious surgical contraindications;
* Expected postoperative survival ≥3 months;
* The study visit plan and other programme requirements are now available;
* Voluntary participation and signing of informed consent.

Exclusion Criteria:

* Patients with stage II and IV periampullary carcinoma of head of pancreas and periampullary carcinoma;
* Active infected persons;
* Distant metastasis or ascites were found in imaging examination;
* Patients with serious impairment of heart, liver and kidney function (grade 3 to 4, ALT and/or AST more than 3 times the normal upper limit, Cr more than the normal upper limit);
* patients with other malignant tumors or blood diseases;
* Pregnancy, planned pregnancy and lactation female patients (urine HCG >02500 iu /L, diagnosed as early pregnancy);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with one or more postoperative complications (time range: 90 days) was observed, and data were recorded during the hospital stay (expected average of 3 weeks) and during control visits 3 months postoperatively. | 3month
  The percentage of patients with one or more postoperative complications (time range: 90 days) was observed, and data were recorded during the hospital stay (expected average of 3 weeks) and during control visits 3 months postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Sahnghai, China